CLINICAL TRIAL: NCT05417022
Title: French Registry to Evaluate the Safety and Efficacy of the Diamondback 360TM Orbital Atherectomy System in the Preparation of Calcified Coronary Lesions Before Implantation of a Coronary Endoprothesis
Brief Title: Safety and Efficacy Evaluation of Orbital Atherectomy System in de Novo Calcified Lesions
Acronym: REFORCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Recherche Cardio Vasculaire Alpes (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02662-39
Record Dates: First submitted 2022-05-13; First posted 2022-06-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Angiography; Coronary Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Diamondback 360TM orbital atherectomy system
  Interventions: Device: Diamondback 360TM orbital atherectomy system

INTERVENTIONS:
Device: Diamondback 360TM orbital atherectomy system — Use of the Diamondback 360TM orbital atherectomy system in the preparation of calcified coronary lesions before implantation of a coronary endoprothesis

SUMMARY:
This is a French, prospective, single-arm, multi-center registry to confirm the safety and efficacy of the Diamondback 360 TM Orbital Atherectomy System in the preparation of de novo calcified coronary lesions before implantation of a coronary endoprothesis in adult subjects. The primary safety endpoint is 30-day MACE and the efficacy endpoint is procedural success.

DETAILED DESCRIPTION:
Treatment of calcified lesions, caused in 6 to 20% of patients, remains a challenge.

Presence of coronary calcifications complicates stent placement resulting in up to 50% malapposition or under-expansion of the stent and is associated with a higher frequency of major adverse cardiac events (MACE).

In order to reduce these risks, preparation of these lesions before the implantation of a coronary stent is essential. The arrival on the European market of a new Orbital atherectomy system leads to consider its use in the preparation of such lesions.

The orbital atherectomy system uses a diamond-coated eccentric crown that abrades calcified plaque and develops pulsatile forces on the wall. It reduces calcified plaque and modifies plaque with fractures, facilitating stent placement and allowing for optimal stent expansion.

ORBIT I and ORBIT II clinical trials were conducted in the United States to evaluate the safety of using the Orbital Atherectomy System in de novo calcified coronary lesions in adults. These 2 trials demonstrated that orbital atherectomy not only facilitated stenting, but also improved clinical outcomes compared to historical outcomes.

The recent obtaining of CE marking allows the use of this very promising medical device in France.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years
* Patients with a clinical indication for coronary angioplasty and presenting a de novo calcified lesion
* The target vessel reference diameter must be >= 2.5mm and <= 4.0 mm.
* Lesion length <= 40 mm
* The target vessel must be a coronary artery with a stenosis of >70%
* Patients able to understand and provide informed consent
* Patients with Social Security coverage

Exclusion Criteria:

* Patients with an LVEF < 25%.
* Patient with hypersensitivity to egg, soy or peanut proteins or to one of the active substances or one of the excipients of ViperSlide lubricant.
* Pregnant or breastfeeding woman
* Unwilling or unable to sign the Informed Consent
* Patients under judicial protection, tutorship or curatorship
* Angiographic criteria: Intra-stent stenosis, Presence of a chronic total occlusion (CTO), Bypass lesion, Target vessel excessively tortuous, Presence of a thrombus, Presence of a single permeable vessel

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who undergo an angioplasty requiring Diamondback 360TM orbital atherectomy System and who agree to participate in this study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint : Major Adverse Cardiac Event (MACE) | 30 days
  The Diamondback 360°® Orbital Atherectomy System safety was evaluated by a composite of MACE at 30-days post procedure. MACE is composed of :
  * Myocardial infarction : Type I and/or Type IV
  * TVR - defined as revascularization at the target vessel after the completion of the index procedure.
  * Cardiac death.

SECONDARY OUTCOMES:
Efficacy Endpoint : Revascularization success rate | Until hospital discharge after index procedure, average estimated at 48 hours
  Revascularization success was defined as successful stent placement with < 30% residual stenosis and without severe angiographic complications during intervention and/or MACE during the period of the patient's hospitalization.
  Severe angiographic complications were defined as severe dissection (Type C to F) , perforation and persistent slow flow or no flow, Atrioventricular conduction disorder.
Safety Endpoint : 12 Month MACE | 12 months
  See MACE definition in the primary outcome.
Safety endpoint : Comparison of MACE with rotational atherectomy | 30 days
  The safety of Orbital Atherectomy System will be compared to rotational atherectomy by comparing the MACE rate at 1 month recorded in this study and that recorded in the Euro4C Study.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Monségu, Principal Investigator — Groupe Hospitalier Mutualiste de Grenoble
Locations (17):
- France (17):
  - GCS-ES Axium-Rambot, Aix-en-Provence
  - Centre Hospitalier Antibes - Juan-Les-Pins, Antibes
  - Hôpital Européen de la Roseraie, Aubervilliers
  - Centre Hospitalier d'Avignon, Avignon
  - Clinique Rhône Durance, Avignon
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Pôle Santé République - ELSAN, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Hospitalier de Haguenau, Haguenau
  - Centre Hospitalier Marne la Vallée, Jossigny
  - Hôpital de la Timone, Marseille
  - Hôpital Privé du Confluent, Nantes
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Clinique Saint Hilaire, Rouen
  - Institut Arnault Tzanck, Saint-Laurent-du-Var
  - CHU Strasbourg, Strasbourg
  - Centre Hospitalier Intercommunal Toulon - La Seyne/Mer, Toulon

REFERENCES:
- [Background] Sturm R, Martinsen BJ, Valle JA, Waldo SW, Behrens AN, Armstrong EJ. Orbital Atherectomy for Treatment of Complex Severely Calcified Coronary Artery Lesions: Insights from a Veterans Affairs Cohort. Cardiovasc Revasc Med. 2020 Mar;21(3):330-333. doi: 10.1016/j.carrev.2019.06.013. Epub 2019 Jun 28. PMID 31307929
- [Background] Mosseri M, Satler LF, Pichard AD, Waksman R. Impact of vessel calcification on outcomes after coronary stenting. Cardiovasc Revasc Med. 2005 Oct-Dec;6(4):147-53. doi: 10.1016/j.carrev.2005.08.008. PMID 16326375
- [Background] Onuma Y, Tanimoto S, Ruygrok P, Neuzner J, Piek JJ, Seth A, Schofer JJ, Richardt G, Wiemer M, Carrie D, Thuesen L, Dorange C, Miquel-Hebert K, Veldhof S, Serruys PW. Efficacy of everolimus eluting stent implantation in patients with calcified coronary culprit lesions: two-year angiographic and three-year clinical results from the SPIRIT II study. Catheter Cardiovasc Interv. 2010 Nov 1;76(5):634-42. doi: 10.1002/ccd.22541. PMID 20690152
- [Background] Fitzgerald PJ, Ports TA, Yock PG. Contribution of localized calcium deposits to dissection after angioplasty. An observational study using intravascular ultrasound. Circulation. 1992 Jul;86(1):64-70. doi: 10.1161/01.cir.86.1.64. PMID 1617791
- [Background] Moussa I, Di Mario C, Moses J, Reimers B, Di Francesco L, Martini G, Tobis J, Colombo A. Coronary stenting after rotational atherectomy in calcified and complex lesions. Angiographic and clinical follow-up results. Circulation. 1997 Jul 1;96(1):128-36. doi: 10.1161/01.cir.96.1.128. PMID 9236427
- [Background] Bhatt P, Parikh P, Patel A, Chag M, Chandarana A, Parikh R, Parikh K. Orbital atherectomy system in treating calcified coronary lesions: 3-Year follow-up in first human use study (ORBIT I trial). Cardiovasc Revasc Med. 2014 Jun;15(4):204-8. doi: 10.1016/j.carrev.2014.03.004. Epub 2014 Mar 19. PMID 24746600
- [Background] Chambers JW, Feldman RL, Himmelstein SI, Bhatheja R, Villa AE, Strickman NE, Shlofmitz RA, Dulas DD, Arab D, Khanna PK, Lee AC, Ghali MG, Shah RR, Davis TP, Kim CY, Tai Z, Patel KC, Puma JA, Makam P, Bertolet BD, Nseir GY. Pivotal trial to evaluate the safety and efficacy of the orbital atherectomy system in treating de novo, severely calcified coronary lesions (ORBIT II). JACC Cardiovasc Interv. 2014 May;7(5):510-8. doi: 10.1016/j.jcin.2014.01.158. PMID 24852804
- [Background] Benezet J, Diaz de la Llera LS, Cubero JM, Villa M, Fernandez-Quero M, Sanchez-Gonzalez A. Drug-eluting stents following rotational atherectomy for heavily calcified coronary lesions: long-term clinical outcomes. J Invasive Cardiol. 2011 Jan;23(1):28-32. PMID 21183767
- [Background] Bouisset F, Barbato E, Reczuch K, Dobrzycki S, Meyer-Gessner M, Bressollette E, Cayla G, Lhermusier T, Zajdel W, Palazuelos Molinero J, Ferenc M, Ribichini FL, Carrie D. Clinical outcomes of PCI with rotational atherectomy: the European multicentre Euro4C registry. EuroIntervention. 2020 Jul 17;16(4):e305-e312. doi: 10.4244/EIJ-D-19-01129. PMID 32250249
- [Background] Kobayashi Y, Okura H, Kume T, Yamada R, Kobayashi Y, Fukuhara K, Koyama T, Nezuo S, Neishi Y, Hayashida A, Kawamoto T, Yoshida K. Impact of target lesion coronary calcification on stent expansion. Circ J. 2014;78(9):2209-14. doi: 10.1253/circj.cj-14-0108. Epub 2014 Jul 14. PMID 25017740
- [Background] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145
- [Background] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Background] Lee M, Genereux P, Shlofmitz R, Phillipson D, Anose BM, Martinsen BJ, Himmelstein SI, Chambers JW. Orbital atherectomy for treating de novo, severely calcified coronary lesions: 3-year results of the pivotal ORBIT II trial. Cardiovasc Revasc Med. 2017 Jun;18(4):261-264. doi: 10.1016/j.carrev.2017.01.011. Epub 2017 Jan 23. PMID 28162989